CLINICAL TRIAL: NCT03825536
Title: Short-term Effects of Methamphetamine Exposure on Residual Viral Transcription During Treated HIV Disease
Brief Title: Effect of Methamphetamine on Residual Latent HIV Disease Study
Acronym: EMRLHD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 18-26765; 1R61DA047024-01 (NIH)
Record Dates: First submitted 2019-01-28; First posted 2019-01-31 (Actual); Results first posted 2025-04-08 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: HIV-1-infection; Methamphetamine-dependence
Keywords: HIV; methamphetamine; viral transcription; inflammation
MeSH Terms: conditions — Inflammation | interventions — Methamphetamine

STUDY DESIGN:
Intervention Model Description: This is a phase IV randomized, double-blinded, placebo-controlled crossover study. A placebo treatment arm will be assigned to participants in a randomized crossover design. HIV+ ART-suppressed individuals with no prior history of MA use disorder will be administered 10mg oral methamphetamine hydrochloride, followed by 15 mg methamphetamine hydrochloride two hours later, for a total of 25mg in one 24-hour period (the maximum FDA approved daily dose for the treatment of childhood obesity). Participants will complete the study twice (once on a placebo treatment arm and once with the oral methamphetamine treatment arm). Which treatment arm occurs first will be randomly assigned and will include a 31-day washout period between the two phases.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The order in which participants complete the two treatment phases (i.e., oral methamphetamine and placebo) will be unknown to both the participants and the PI/study team. Both the oral methamphetamine and placebo will be prepared in identical capsules by the UCSF investigational pharmacist, out of sight of the study participant, study coordinator, and study site PI and administered to the participant to maintain double blinding. The investigational pharmacist will randomize each participant according to the methods described above. In the event that participant experiences an adverse event that requires the identity of the study drug be revealed, the PI will be able to contact the investigational pharmacist to break the blind. In the event that a participant blind is broken, the study PIs will determine the impact upon the un-blinded participant's continued participation in the study and if a replacement participant is needed on a case-by-case basis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral methamphetamine, then Placebo oral capsule (Experimental): Participants will be randomized to oral methamphetamine first then placebo oral capsule using a random number generator. When oral methamphetamine is administered, an initial 10 mg of oral methamphetamine study drug will be administered to assess tolerability, followed by a subsequent 15 mg oral dose two hours later. Then the participant will receive the placebo oral capsule for their second treatment phase starting at approximately Day 77. For the placebo treatment, one placebo capsule will be administered orally on treatment day, followed by a second oral placebo capsule two hours later.
  Interventions: Drug: Oral Methamphetamine; Other: Placebo oral capsule
- Placebo oral capsule, then Oral methamphetamine (Experimental): Participants will be randomized to a placebo oral capsule first, then oral methamphetamine using a random number generator. For the placebo treatment, one placebo capsule will be administered orally on treatment day, followed by a second oral placebo capsule two hours later. Then the participant will receive the oral methamphetamine capsule for their second treatment phase starting at approximately Day 77. When oral methamphetamine is administered, an initial 10 mg of oral methamphetamine study drug will be administered to assess tolerability, followed by a subsequent 15 mg oral dose two hours later.
  Interventions: Drug: Oral Methamphetamine; Other: Placebo oral capsule

INTERVENTIONS:
Drug: Oral Methamphetamine — An initial 10 mg of oral methamphetamine (over-encapsulated to look similar to placebo capsule) study drug will be administered to assess tolerability, followed by a subsequent 15 mg oral dose (over-encapsulated to look similar to placebo capsule) two hours later.
  Other Names: Desoxyn
Other: Placebo oral capsule — One placebo capsule will be administered orally on treatment day, followed by a second oral placebo capsule two hours later.
  Other Names: Placebo

SUMMARY:
The most commonly used illicit stimulant in HIV-infected individuals is methamphetamine (MA). Prior studies demonstrate strong evidence that MA promotes increased HIV transcription as well as immune dysregulation. A challenge in achieving worldwide HIV eradication is targeting specific marginalized populations who are most likely to benefit from an HIV cure but possess poorer immune responses. For this study, HIV+ infected ART-suppressed individuals with no prior history of MA use disorder will be administered oral methamphetamine (the maximum FDA approved daily dose for the treatment of childhood obesity) to determine the effects of short-term MA exposure on residual virus production, gene expression, and inflammation. Measures of MA exposure in urine and serum will then be associated with residual virus production, gene expression, cell surface immune marker protein expression, and systemic markers of inflammation. The clinical trial data will generate advanced gene expression and immunologic data to identify potential novel targets for reversing HIV latency, reducing inflammation, and personalizing future therapies in HIV+ individuals who use MA.

DETAILED DESCRIPTION:
The most commonly used illicit stimulant in HIV-infected individuals is methamphetamine (MA), and prior studies demonstrate strong evidence that MA promotes increased HIV transcription as well as immune dysregulation. HIV cure has emerged as an important clinical and research priority given evidence of ongoing immune dysfunction in HIV-infected individuals despite effective antiretroviral therapy (ART). A challenge in achieving worldwide HIV eradication is targeting specific vulnerable populations who are most likely to benefit from an HIV cure but possess poorer immune responses as a result of residual viral replication due to suboptimal ART adherence and/or direct immune dysfunction from illicit substance use. Prior non-human studies demonstrate that MA directly induces HIV production and promotes immune activation and inflammation. These preclinical findings suggest that HIV+ individuals who use MA may experience greater immune dysfunction and face additional challenges for future HIV eradication. This study will investigate the effects of short-term MA exposure in HIV+ ART-suppressed individuals without a prior history of MA use. Participants will be enrolled in an interventional study where they will be administered oral methamphetamine (the maximum FDA approved daily dose for the treatment of childhood obesity) to determine the effects of short-term MA exposure on residual virus production, gene expression, inflammation, and trace amine-associated 1 (TAAR1, a promising drug target for psychostimulant addiction) signaling. MA exposure will be quantified with multiple serum samples collected over a 24-hour monitoring period and associated with residual viral transcription, host gene and cell surface protein expression, and inflammation (plasma inflammatory cytokine levels) quantification. The proposed study will be the first human genetic study to directly evaluate the effect of MA exposure on residual viral transcription during effective ART. The overall goals of the study are to integrate a rigorous clinical study designs with high throughput 'omics data to identify novel targets for reversing HIV latency, reducing inflammation, and personalizing future therapeutic strategies specific to HIV+ ART-suppressed individuals who use MA.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent
2. Male or female, age ≥ 18 and ≤ 65 years
3. HIV-1 infection, documented by any licensed rapid HIV test or HIV enzyme or chemiluminescence immunoassay (E/CIA) test kit at any time prior to study entry and confirmed by a licensed Western blot or a second antibody test by a method other than the initial rapid HIV and/or E/CIA, or by HIV-1 antigen or plasma HIV-1 RNA viral load.
4. Continuous therapy with a Department of Health and Human Services (DHHS) recommended/alternative combination ART for least 24 months (at least 3 agents) at study entry with no regimen changes in the preceding 12 weeks
5. Maintenance of undetectable plasma HIV-1 RNA (<40 copies/ml) for at least 12 months. Episodes of single HIV plasma RNA 50-500 copies/ml will not exclude participation if subsequent HIV plasma RNA is <40 copies/ml.
6. No plans to modify ART during the study period (146 days, or approximately 5 months)
7. Screening CD4+ (cluster of differentiation 4) T-cell count ≥ 350 cells/mm3
8. Screening hemoglobin ≥ 12.5 g/dL
9. No current or prior history of methamphetamine (MA) use disorder by DSM-5 diagnostic criteria. Participants may have a prior history of taking prescription medications containing amphetamines-type stimulants such as Adderall® or Dexedrine® or Ritalin for the treatment of conditions such as attention deficit hyperactivity disorder as long as the participant has not taken these medications in the last 12 months or plans to take these medications during the entire study period.
10. Willingness to use two forms of contraception throughout the study period as well as up to 30 days after the last day of study completion.
11. Ability and availability to participate in the full 146 days of the study (approximately 5 month) and maintain the inclusion/exclusion criteria.

Exclusion Criteria:

1. History of methamphetamine ("meth") use disorder by DSM-5 diagnostic criteria.
2. Evidence of MA use other than due to the administered oral methamphetamine study drug, based on urine, hair, or serum MA measurements collected at baseline and follow-up study visits.
3. Current use of prescription medications containing amphetamine-type stimulants (e.g., Adderall®, Dexedrine®, Ritalin, etc.) within the last 1 year.
4. Sensitivity or allergy to amphetamine-type stimulants
5. Current use of any other "psychoactive" drug within the last 1 year. These include cocaine, ecstasy, lysergic acid diethylamide (LSD), mushrooms, or other recreational drugs - but nicotine or caffeine use is ok.
6. Marijuana use in the last 30 days; marijuana may influence the interpretation of the study drug's effect on viral transcription, inflammation, and/or gene expression.
7. Current use of opioids (heroin, methadone) or prescription opioid agonists such as hydrocodone (Norco®), buprenorphine/naloxone (Suboxone®), oxycodone (Oxycontin®), hydromorphone (Dilaudid®) within the last 1 year by self-report and/or urine qualitative screening.
8. Current use of alcohol use disorder (DSM-5 criteria) within the last 1 year as this might put patient at risk of withdrawal during the study.
9. Significant physical or psychiatric illness that might impair the ability to safely complete the study or that might be complicated by the study drugs, including prior seizures (after age 8) or other active neurological disease.
10. Clinically significant abnormalities on physical examination or screening laboratory values
11. History of serious adverse event or hypersensitivity to MA or corn starch (the latter is used in the placebo).
12. Recent use within the last month of the following medications given potential interactions with oral methamphetamine: acebrophylline, iobenguane, isocarboxazid, methylene blue, moclobemide, phenelzine, procarbazine, rasagiline, safinamide, selegiline, tranylcypromine, asunaprevir, buproprion, topical cocaine, fluoxetine, iohexol, linezolid, paroxetine, potassium citrate, quinidine, sodium bicarbonate, sodium citrate, sodium lactate, tipranavir, and tromethamine.
13. Recent hospitalization in the last 90 days.
14. Recent infection in the last 90 days requiring systemic antibiotics.
15. Screening hemoglobin below 12.5 g/dL.
16. Prior diagnosis or abnormal screening labs consistent with a diagnosis of hyperthyroidism or hypothyroidism.
17. Poorly controlled hypertension with systolic blood pressure > 160 on more than one occasion.
18. History of glaucoma.
19. Significant myocardial disease (current myocarditis or reduced left ventricular ejection fraction below the lower limit of normal) or diagnosed coronary artery disease.
20. History of psychotic symptoms (e.g., hallucinations, delusional thinking).
21. History of bipolar disorder.
22. Significant respiratory disease requiring oxygen.
23. A history of hypersensitivity to sympathomimetic amines (e.g., epinephrine, norepinephrine, or dopamine).
24. Diabetes or current hypothyroidism.
25. Participants of reproductive potential or breastfeeding. Women of childbearing potential must have a negative serum pregnancy test at screening. All participants of childbearing potential must agree to use a double-barrier method of contraception throughout the study period and up to 90 days after the last dose of MA.
26. Exposure to any immunomodulatory drug (including maraviroc) in the 16 weeks prior to study.
27. Prior or current use of experimental agents used with the intent to perturb the HIV-1 viral reservoir.
28. History of seizures, psychosis, abnormal electroencephalogram or brain damage with significant persisting neurological deficit
29. Recent vaccination within the last 2 weeks prior to study baseline visit. Routine or standard of care vaccinations (such as influenza, pneumococcal, and meningococcal vaccinations) are allowed but must be administered greater than 14 days prior to baseline study visit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-01-11 (Actual); Study Completion 2023-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sulggi A Lee, MD PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco General Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Castillo-Mancilla JR, Brown TT, Erlandson KM, Palella FJ Jr, Gardner EM, Macatangay BJ, Breen EC, Jacobson LP, Anderson PL, Wada NI. Suboptimal Adherence to Combination Antiretroviral Therapy Is Associated With Higher Levels of Inflammation Despite HIV Suppression. Clin Infect Dis. 2016 Dec 15;63(12):1661-1667. doi: 10.1093/cid/ciw650. Epub 2016 Sep 22. PMID 27660234
- [Background] Passaro RC, Pandhare J, Qian HZ, Dash C. The Complex Interaction Between Methamphetamine Abuse and HIV-1 Pathogenesis. J Neuroimmune Pharmacol. 2015 Sep;10(3):477-86. doi: 10.1007/s11481-015-9604-2. Epub 2015 Apr 8. PMID 25850893
- [Background] Centers for Disease Control and Prevention (CDC). Increasing morbidity and mortality associated with abuse of methamphetamine--United States, 1991-1994. MMWR Morb Mortal Wkly Rep. 1995 Dec 1;44(47):882-6. PMID 7476843
- [Background] Marquez C, Mitchell SJ, Hare CB, John M, Klausner JD. Methamphetamine use, sexual activity, patient-provider communication, and medication adherence among HIV-infected patients in care, San Francisco 2004-2006. AIDS Care. 2009 May;21(5):575-82. doi: 10.1080/09540120802385579. PMID 19444665
- [Background] Wires ES, Alvarez D, Dobrowolski C, Wang Y, Morales M, Karn J, Harvey BK. Methamphetamine activates nuclear factor kappa-light-chain-enhancer of activated B cells (NF-kappaB) and induces human immunodeficiency virus (HIV) transcription in human microglial cells. J Neurovirol. 2012 Oct;18(5):400-10. doi: 10.1007/s13365-012-0103-4. Epub 2012 May 22. PMID 22618514
- [Background] Liang H, Wang X, Chen H, Song L, Ye L, Wang SH, Wang YJ, Zhou L, Ho WZ. Methamphetamine enhances HIV infection of macrophages. Am J Pathol. 2008 Jun;172(6):1617-24. doi: 10.2353/ajpath.2008.070971. Epub 2008 May 5. PMID 18458095
- [Background] Toussi SS, Joseph A, Zheng JH, Dutta M, Santambrogio L, Goldstein H. Short communication: Methamphetamine treatment increases in vitro and in vivo HIV replication. AIDS Res Hum Retroviruses. 2009 Nov;25(11):1117-21. doi: 10.1089/aid.2008.0282. PMID 19895343
- [Background] Jiang J, Wang M, Liang B, Shi Y, Su Q, Chen H, Huang J, Su J, Pan P, Li Y, Wang H, Chen R, Liu J, Zhao F, Ye L, Liang H. In vivo effects of methamphetamine on HIV-1 replication: A population-based study. Drug Alcohol Depend. 2016 Feb 1;159:246-54. doi: 10.1016/j.drugalcdep.2015.12.027. Epub 2016 Jan 4. PMID 26790825
- [Background] Saito M, Yamaguchi T, Kawata T, Ito H, Kanai T, Terada M, Yokosuka M, Saito TR. Effects of methamphetamine on cortisone concentration, NK cell activity and mitogen response of T-lymphocytes in female cynomolgus monkeys. Exp Anim. 2006 Oct;55(5):477-81. doi: 10.1538/expanim.55.477. PMID 17090965
- [Background] Harms R, Morsey B, Boyer CW, Fox HS, Sarvetnick N. Methamphetamine administration targets multiple immune subsets and induces phenotypic alterations suggestive of immunosuppression. PLoS One. 2012;7(12):e49897. doi: 10.1371/journal.pone.0049897. Epub 2012 Dec 5. PMID 23227154
- [Background] Carrico AW, Flentje A, Kober K, Lee S, Hunt P, Riley ED, Shoptaw S, Flowers E, Dilworth SE, Pahwa S, Aouizerat BE. Recent stimulant use and leukocyte gene expression in methamphetamine users with treated HIV infection. Brain Behav Immun. 2018 Jul;71:108-115. doi: 10.1016/j.bbi.2018.04.004. Epub 2018 Apr 18. PMID 29679637
- [Background] Jing L, Li JX. Trace amine-associated receptor 1: A promising target for the treatment of psychostimulant addiction. Eur J Pharmacol. 2015 Aug 15;761:345-52. doi: 10.1016/j.ejphar.2015.06.019. Epub 2015 Jun 16. PMID 26092759
- [Background] Pei Y, Asif-Malik A, Hoener M, Canales JJ. A partial trace amine-associated receptor 1 agonist exhibits properties consistent with a methamphetamine substitution treatment. Addict Biol. 2017 Sep;22(5):1246-1256. doi: 10.1111/adb.12410. Epub 2016 May 19. PMID 27193165
- [Background] Panas MW, Xie Z, Panas HN, Hoener MC, Vallender EJ, Miller GM. Trace amine associated receptor 1 signaling in activated lymphocytes. J Neuroimmune Pharmacol. 2012 Dec;7(4):866-76. doi: 10.1007/s11481-011-9321-4. Epub 2011 Oct 29. PMID 22038157
- [Background] Uhl GR, Drgon T, Liu QR, Johnson C, Walther D, Komiyama T, Harano M, Sekine Y, Inada T, Ozaki N, Iyo M, Iwata N, Yamada M, Sora I, Chen CK, Liu HC, Ujike H, Lin SK. Genome-wide association for methamphetamine dependence: convergent results from 2 samples. Arch Gen Psychiatry. 2008 Mar;65(3):345-55. doi: 10.1001/archpsyc.65.3.345. PMID 18316681
- [Background] Breen MS, Uhlmann A, Nday CM, Glatt SJ, Mitt M, Metsalpu A, Stein DJ, Illing N. Candidate gene networks and blood biomarkers of methamphetamine-associated psychosis: an integrative RNA-sequencing report. Transl Psychiatry. 2016 May 10;6(5):e802. doi: 10.1038/tp.2016.67. PMID 27163203
- [Background] Li MD, Wang J, Niu T, Ma JZ, Seneviratne C, Ait-Daoud N, Saadvandi J, Morris R, Weiss D, Campbell J, Haning W, Mawhinney DJ, Weis D, McCann M, Stock C, Kahn R, Iturriaga E, Yu E, Elkashef A, Johnson BA. Transcriptome profiling and pathway analysis of genes expressed differentially in participants with or without a positive response to topiramate treatment for methamphetamine addiction. BMC Med Genomics. 2014 Dec 12;7:65. doi: 10.1186/s12920-014-0065-x. PMID 25495887

RESULTS

PARTICIPANT FLOW:
Period: First Intervention (30 Days)
Arm/Group | Oral Methamphetamine, Then Placebo Oral Capsule | Placebo Oral Capsule, Then Oral Methamphetamine
Started | 7 | 7
Completed | 5 | 6
Not Completed | 2 | 1
Period: Washout (30 Days)
Arm/Group | Oral Methamphetamine, Then Placebo Oral Capsule | Placebo Oral Capsule, Then Oral Methamphetamine
Started | 5 | 6
Completed | 5 | 5
Not Completed | 0 | 1
Period: Second Intervention (30 Days)
Arm/Group | Oral Methamphetamine, Then Placebo Oral Capsule | Placebo Oral Capsule, Then Oral Methamphetamine
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Methamphetamine, Then Placebo Oral Capsule | Placebo Oral Capsule, Then Oral Methamphetamine | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.6 (9.50) | 44.4 (9.34) | 45 (8.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 5 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 4 | 3 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 3 | 5 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: HIV Transcription (Cell-associated HIV RNA) in Peripheral Blood
Description: The change in HIV reservoir size (as measured by cell-associated HIV RNA levels) over a 4 hour study period.
Time Frame: 4 hours
Measure: Median (Inter-Quartile Range); unit: copies/million cells
Arm/Group | Oral Methamphetamine, Then Placebo Oral Capsule | Placebo Oral Capsule, Then Oral Methamphetamine
Number analyzed (Participants) | 5 | 5
copies/million cells | 10.45 [1.3 to 31.79] | 57.38 [27.59 to 404.7]

2. Secondary Outcome: Systemic Inflammation (Plasma Pro-inflammatory Cytokine Levels)
Description: The change in plasma pro-inflammatory IL-1B levels over a 4 hour study period.
Time Frame: 4 hours
Measure: Median (Inter-Quartile Range); unit: pg/uL
Groups:
- Oral Methamphetamine: An initial 10 mg of oral methamphetamine (over-encapsulated to look similar to placebo capsule) study drug was administered to assess tolerability, followed by a subsequent 15 mg oral dose (over-encapsulated to look similar to placebo capsule) two hours later.
- Placebo Oral Capsule: One placebo oral capsule was administered orally on treatment day, followed by a second oral placebo capsule two hours later.
Arm/Group | Oral Methamphetamine | Placebo Oral Capsule
Number analyzed (Participants) | 10 | 10
pg/uL | 0.875 [0.000 to 3.473] | 0.054 [-0.032 to 0.560]

3. Secondary Outcome: Host Gene Expression (RNA Sequencing) in Peripheral Blood
Description: The change in host gene expression as measured by RNA-seq over a 4 hour study period
Time Frame: 4 hours
Reporting Status: Not Posted

4. Secondary Outcome: Trace Amine Receptor 1 (TAAR1) Signaling Metabolite Levels in in Peripheral Blood
Description: The change in tyramine (TAAR1 signaling metabolite) levels over a 4 hour study period.
Time Frame: 4 hours
Measure: Median (Inter-Quartile Range); unit: ug
Arm/Group | Oral Methamphetamine | Placebo Oral Capsule
Number analyzed (Participants) | 9 | 9
ug | -215.901 [-296.094 to -132.644] | -171.506 [-340.327 to -92.9]

ADVERSE EVENTS:
Time Frame: 4 months
Description: Regular monitoring of vitals (e.g. BP, O2 levels) and ECG by MD present before and after administration of dosages on treatment days.
Arm/Group | Oral Methamphetamine | Placebo Oral Capsule
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 1/14 | 0/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Methamphetamine (N=14) | Placebo Oral Capsule (N=14)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-20): https://cdn.clinicaltrials.gov/large-docs/36/NCT03825536/Prot_SAP_000.pdf
  • Informed Consent Form (2022-02-03): https://cdn.clinicaltrials.gov/large-docs/36/NCT03825536/ICF_001.pdf